CLINICAL TRIAL: NCT03659916
Title: An Open-label Extension Study to Evaluate Long-term Efficacy and Safety of A4250 in Children With Progressive Familial Intrahepatic Cholestasis Types 1 and 2 (PEDFIC 2)
Brief Title: Long Term Safety & Efficacy Study Evaluating The Effect of A4250 in Children With PFIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo, an Ipsen Company (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250-008; 2017-002325-38 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-09-06 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
Keywords: Pediatric; Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis | interventions — odevixibat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A4250 (Experimental): Capsules for oral administration (40 or 120 µg/kg) once daily for 72 weeks, or 40 µg/kg/day for the first 12 weeks followed by 120 µg/kg/day for the remaining 60 weeks"
  Interventions: Drug: A4250 (odevixibat)

INTERVENTIONS:
Drug: A4250 (odevixibat) — A4250 is a small molecule and selective inhibitor of IBAT

SUMMARY:
Open Label Extension Study to evaluate long term safety and persistence of effect of A4250 in children with PFIC.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

1. Completion of the 24-week Treatment Period of Study A4250-005 or withdrawn from Study A4250-005 due to patient/caregiver judgment of intolerable symptoms after completing at least 12 weeks of treatment
2. Signed informed consent and assent as appropriate
3. Patients expected to have a consistent caregiver for the duration of the study
4. Caregivers (and age appropriate patients) must be willing and able to use an eDiary device as required by the study

Inclusion Criteria Cohort 2:

1. A male or female patient of any age, with a clinical diagnosis of PFIC, including episodic forms (i.e., BRIC), and with a body weight ≥5 kg at Visit S-1.
2. Patient must have clinical genetic confirmation of PFIC
3. Patients with PFIC, excluding BRIC, must have elevated serum bile acid concentration,specifically measured to be ≥100 μmol/L, taken as the average of 2 samples at least 7 days apart (Visits S-1 and S-2) prior to the Screening/Inclusion Visit (Visit 1).
4. Patients with PFIC, excluding BRIC, must have history of significant pruritus and a caregiver-reported observed scratching or patient-reported itching (for patients >18 with no caregiver-reported observed scratching) in the eDiary average of ≥2 (on 0 to 4 scale) in the 2 weeks prior to the Screening/Inclusion Visit (Visit 1).
5. Patients with episodic forms of PFIC (i.e., BRIC) must have an emerging flare characterized by clinically significant pruritus and elevated serum bile acid levels/cholestasis as judged by the investigator.
6. Patient and/or legal guardian must sign informed consent (and assent) as appropriate. Patients who turn 18 years of age (or legal age per country) during the study will be required to re-consent in order to remain in the study.
7. Age appropriate patients are expected to have a consistent caregiver for the duration of the study
8. Caregivers and age-appropriate patients (≥8 years of age) must be willing and able to use an eDiary device as required by the study

Exclusion Criteria Cohort 1:

1. Decompensated liver disease: coagulopathy, history, or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy
2. Sexually active males and females who are not using a reliable contraceptive method with ≤1% failure rate (such as hormonal contraception, intra-uterine device, or complete abstinence) throughout the duration of the study and 90 days thereafter
3. Patients not compliant with treatment in study A4250-005
4. Any other conditions or abnormalities which, in the opinion of the investigator or Medical Monitor, may compromise the safety of the patient, or interfere with the patient participating in or completing the study

Exclusion Criteria Cohort 2:

1. Known pathologic variations of the ABCB11 gene that have been demonstrated to result in complete absence of the BSEP protein
2. Patient with past medical history or ongoing presence of other types of liver disease including, but not limited to, the following:

   1. Biliary atresia of any kind
   2. Suspected or proven liver cancer or metastasis to the liver on imaging studies
   3. Histopathology on liver biopsy is suggestive of alternate non-PFIC related etiology of cholestasis Note: Patients with clinically significant portal hypertension are allowed.
3. Patient with a past medical history or ongoing presence of any other disease or condition known to interfere with the absorption, distribution, metabolism (specifically bile acid metabolism), or excretion of drugs in the intestine, including but not limited to,inflammatory bowel disease.
4. Patient with past medical history or ongoing chronic (i.e., >3 months) diarrhea requiring intravenous fluid or nutritional intervention for treatment of the diarrhea and/or its sequelae.
5. Patient has a confirmed past diagnosis of infection with human immunodeficiency virus or other present and active, clinically significant, acute, or chronic infection, or past medical history of any major episode of infection requiring hospitalization or treatment with parenteral anti-infective treatment within 4 weeks of treatment start (Study Day 1) or completion of oral anti-infective treatment within 2 weeks prior to start of Screening Period.
6. Any patient with suspected or confirmed cancers except for basal cell carcinoma, and non-liver cancers treated at least 5 years prior to Screening with no evidence of recurrence.
7. Patient has had a liver transplant, or a liver transplant is planned within 6 months of the Screening/Inclusion Visit.
8. Decompensated liver disease, coagulopathy, history, or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy
9. INR >1.4 (the patient may be treated with Vitamin K intravenously, and if INR is ≤1.4 at resampling the patient may be included).
10. Serum ALT >10 × upper limit of normal (ULN) at Screening.
11. Serum ALT >15 × ULN at any time point during the last 6 months unless an alternate etiology was confirmed for the elevation.
12. Total bilirubin >10 × ULN at Screening.
13. Patient suffers from uncontrolled, recalcitrant pruritic condition other than PFIC.

    Examples include, but not limited to, refractory atopic dermatitis or other primary pruritic skin diseases.
14. Any patient who is pregnant or lactating or who is planning to become pregnant within 72 weeks of the Screening/Inclusion Visit.
15. Sexually active males and females who are not using a reliable contraceptive method with ≤1% failure rate (such as hormonal contraception, intrauterine device, or complete abstinence) throughout the duration of the study and 90 days thereafter (from signed informed consent through 90 days after last dose of study drug).
16. Patient with a past medical history of alcohol or substance abuse will be excluded. Patient must agree to refrain from illicit drug and alcohol use during the study.
17. Administration of bile acid or lipid binding resins and medications that slow GI motility.
18. Patient has had investigational exposure to a drug, biologic agent, or medical device within 30 days prior to Screening, or 5 half-lives of the study agent, whichever is longer.
19. Any other conditions or abnormalities which, in the opinion of the investigator or Medical Monitor, may compromise the safety of the patient, or interfere with the patient participating in or completing the study.

Ages: 0 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2025-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (41):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Riley Hospital for Children - Riley Children's Specialists, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center - Presbyterian Hospital Building, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine - Texas Children's Liver Center, Houston, Texas
- The Royal Children's Hospital, Melbourne, Australia
- Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Belgium
- The Hospital for Sick Children, Toronto, Canada
- France (4):
  - University and Pediatric Hospital of Lyon, Bron
  - Universite Paris SUD - Hpitaux Universitaires Paris-Sud - Hopital Bicetre, Le Kremlin-Bicêtre
  - Hospital De La Timone, Marseille
  - Hospital Necker-Enfants Maladies, Paris
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Kinderklinik Tubingen, Universitatsklinikum Tubingen, Tübingen
  - Univesitatsklinikum Tubingen Klinik fur Kinder und Jugendmedizin, Tübingen
- Israel (2):
  - Shaare-Zedek Mc, Jerusalem
  - Schneider Children's Medical Center Of Israel, Petah Tikva
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - University Hospital Of Padova, Padua
  - Ospedale Regina Margherita, Torino
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Universitair Medisch Centrum (UMC) Utrecht, Utrecht
- Instytut Pomnik - Centrum Zarowia Dziecka, Warsaw, Poland
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Astrid Lindgren Children's Hospital, Karolinska University Hospital, Solna, Sweden
- Turkey (Türkiye) (5):
  - Gazi University, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Akdeniz University, Antalya
  - Istanbul University Medical Faculty, Istanbul
  - Inonu University Medical Faculty, Malatya
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Leeds General Infirmary, Leeds
  - Institute of Liver Studies - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers

REFERENCES:
- [Derived] Thompson RJ, Artan R, Baumann U, Calvo PL, Czubkowski P, Dalgic B, D'Antiga L, Di Giorgio A, Durmaz O, Gonzales E, Grammatikopoulos T, Gupte G, Hardikar W, Houwen RHJ, Kamath BM, Karpen SJ, Lacaille F, Lachaux A, Lainka E, Loomes KM, Mack CL, Mattsson JP, McKiernan P, Ni Q, Ozen H, Rajwal SR, Roquelaure B, Shteyer E, Sokal E, Sokol RJ, Soufi N, Sturm E, Tessier ME, van der Woerd WL, Verkade HJ, Vittorio JM, Wallefors T, Warholic N, Yu Q, Horn P, Kjems L. Interim results from an ongoing, open-label, single-arm trial of odevixibat in progressive familial intrahepatic cholestasis. JHEP Rep. 2023 Apr 29;5(8):100782. doi: 10.1016/j.jhepr.2023.100782. eCollection 2023 Aug. PMID 37456676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, open-label extension was conducted in participants with progressive familial intrahepatic cholestasis (PFIC) at 43 centers in 13 countries (Belgium, France, Germany, Italy, Netherlands, Poland, United Kingdom, United States [US], Australia, Canada, Israel, Saudi Arabia, and Turkey). The first participant was enrolled on 28 September 2018 and data cut-off (DCO) date was 15 February 2024.
Pre-assignment Details: This study consisted of a 72-week treatment period and a 4-week follow-up period. An optional extension period for continued treatment until commercial availability of odevixibat followed the 72-week treatment period. A total of 116 participants were enrolled in the study. Results are presented up to DCO of 15 February 2024.
Groups:
- Cohort 1: Placebo/Odevixibat: Participants who previously received placebo in study A4250-005 (NCT03566238) for 24 weeks received odevixibat capsule orally at a dose of 120 microgram/kilogram/day (mcg/kg/day) for 72 weeks, unless they required down-titration to the 40 mcg/kg/day due to tolerability issues.
- Cohort 1: Odevixibat/Odevixibat: Participants who previously received odevixibat capsule orally at a dose of 40 or 120 mcg/kg/day in study A4250-005 (NCT03566238) for 24 weeks received odevixibat capsule orally at a dose of 120 mcg/kg/day for 72 weeks, unless they required down-titration to the 40 mcg/kg/day due to tolerability issues.
- Cohort 2: Odevixibat: Participants any age with any type of PFIC who either did not meet eligibility criteria for study A4250-005 (NCT03566238) or were eligible for enrolment in A4250-005 (NCT03566238) after recruitment was complete received odevixibat at a dose of 120 μg/kg/day or following protocol amendment 6.0, initiated at a dose of 40 mcg/kg/day with the possibility to dose escalate to 120 mcg/kg/day after 12 weeks if there was no improvement in pruritus based on investigator judgement, up to 72 weeks.
Period: Treatment Period (72 Weeks)
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Started | 19 | 37 | 60
Completed | 15 | 28 | 40
Not Completed | 4 | 9 | 20
Not completed — Adverse Event | 2 | 1 | 6
Not completed — Withdrawal by Subject | 1 | 4 | 4
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 1 | 3 | 9
Period: Optional Extension Treatment (176 Weeks)
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Started | 14 (1 participant did not enter Optional Extension treatment) | 27 (1 participant did not enter Optional Extension treatment) | 33 (7 participants did not enter Optional Extension treatment)
Completed | 0 | 0 | 0
Not Completed | 14 | 27 | 33
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Transition to Commercial Drug | 5 | 17 | 11
Not completed — Other | 4 | 0 | 3
Not completed — Ongoing Optional Extension Period | 5 | 9 | 17

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all participants who received at least 1 dose of study treatment.
Groups:
- Cohort 1: Placebo/Odevixibat: Participants who previously received placebo in study A4250-005 (NCT03566238) for 24 weeks received odevixibat capsule orally at a dose of 120 mcg/kg/day for 72 weeks, unless they required down-titration to the 40 mcg/kg/day due to tolerability issues.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat | Total
Number analyzed (Participants) | 19 | 37 | 60 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.34 (3.962) | 4.75 (3.711) | 7.62 (7.208) | 6.17 (5.977)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 25 | 52
  Male | 12 | 17 | 35 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 18 | 37 | 50 | 105
  Unknown or Not Reported | 0 | 0 | 8 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 31 | 53 | 100
  Black/African American | 0 | 1 | 2 | 3
  Asian | 2 | 3 | 2 | 7
  Other | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Bile Acids
Description: Blood samples for analysis of fasting total serum bile acids were drawn at specified timepoints. Participants were to fast (water intake only) for at least 4 hours prior to the collection of samples for serum bile acids. Exceptions were made for infants <12 months of age if unable to fast for the full 4 hours. Baseline for Cohort 1 placebo/odevixibat and Cohort 2 groups was defined as the average of last 2 values before the first dose of study treatment in the study. Baseline for Cohort 1 odevixibat/odevixibat group was defined as average of last 2 values before the first dose of study treatment in study A4250-005 (NCT03566238).
Time Frame: Baseline and Week 72
Population: The FAS consisted of all participants who had received at least 1 dose of the study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: micromole per liter (µmol/L)
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 15 | 28 | 43
micromole per liter (µmol/L) | -104.00 (167.318) | -139.84 (172.070) | -57.97 (137.990)

2. Primary Outcome: Proportion of Positive Pruritus Assessments at the Participant Level Over 72-Week Using the Albireo Observer-Reported Outcome (ObsRo) Instrument
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least a 1-point drop from baseline on the Albireo ObsRO instrument. The proportion of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant.
Time Frame: Baseline and Week 72
Population: The FAS consisted of all participants who had received at least 1 dose of the study treatment. Only participants with data collected at Baseline and Week 72 are reported.
Measure: Mean (Standard Deviation); unit: proportion of pruritus-participant-level
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 12 | 26 | 31
proportion of pruritus-participant-level | 55.20 (38.733) | 38.58 (34.877) | 77.28 (28.084)

3. Secondary Outcome: Proportion of Positive Pruritus Assessments at the Participant Level Using the Albireo ObsRo Instrument From Weeks 0-4, 0-12, 0-22, 0-24, 0-36, 0-46, 0-48, 0-60, and 0-70
Description: as for outcome 2
Time Frame: Weeks 0-4, Weeks 0-12, Weeks 0-22, Weeks 0-24, Weeks 0-36, Weeks 0-46, Weeks 0-48, Weeks 0-60, and Weeks 0-70
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of pruritus-participant-level
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 37 | 53
proportion of pruritus-participant-level
  Weeks 0 - 4 | 45.72 (34.300) | 23.64 (27.005) | 60.14 (33.985)
  Weeks 0 - 12: number analyzed (Participants) | 19 | 37 | 50
  Weeks 0 - 12 | 51.05 (37.670) | 27.34 (28.687) | 67.63 (33.645)
  Weeks 0 - 22: number analyzed (Participants) | 17 | 36 | 48
  Weeks 0 - 22 | 56.01 (38.537) | 31.09 (31.859) | 70.05 (33.858)
  Weeks 0 - 24: number analyzed (Participants) | 17 | 36 | 45
  Weeks 0 - 24 | 56.00 (38.331) | 31.45 (32.324) | 68.55 (34.116)
  Weeks 0 - 36: number analyzed (Participants) | 16 | 31 | 43
  Weeks 0 - 36 | 54.63 (38.243) | 33.66 (33.704) | 69.97 (33.872)
  Weeks 0 - 46: number analyzed (Participants) | 14 | 28 | 37
  Weeks 0 - 46 | 60.41 (39.491) | 34.70 (35.593) | 75.46 (29.801)
  Weeks 0 - 48: number analyzed (Participants) | 14 | 29 | 41
  Weeks 0 - 48 | 61.61 (39.936) | 33.56 (35.668) | 74.79 (30.843)
  Weeks 0 - 60: number analyzed (Participants) | 13 | 31 | 35
  Weeks 0 - 60 | 57.80 (38.873) | 33.18 (34.935) | 74.89 (30.434)
  Weeks 0 - 70: number analyzed (Participants) | 13 | 22 | 29
  Weeks 0 - 70 | 58.18 (38.766) | 40.59 (34.928) | 75.60 (29.514)

4. Secondary Outcome: Change From Baseline in Serum Bile Acids at Weeks 4, 12, 22, 24, 36, 46, 48, 60, 70, and 72
Description: Blood samples for analysis of fasting total serum bile acids were drawn at specified timepoints. Participants were to fast (water intake only) for at least 4 hours prior to the collection of samples for serum bile acids. Exceptions were made for infants <12 months of age if unable to fast for the full 4 hours. Baseline for Cohort 1 placebo/odevixibat, and Cohort 2 groups was defined as the average of last 2 values before the first dose of study treatment in the study. Baseline for Cohort 1 odevixibat/odevixibat group was defined as average of last 2 values before the first dose of study treatment in study A4250-005 (NCT03566238).
Time Frame: Baseline and Weeks 4, 12, 22, 24, 36, 46, 48, 60, 70, and 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 18 | 35 | 54
µmol/L
  Week 4: number analyzed (Participants) | 17 | 34 | 53
  Week 4 | -115.76 (151.014) | -118.78 (172.353) | -76.92 (94.662)
  Week 12 | -98.39 (149.118) | -109.90 (176.472) | -65.01 (136.303)
  Week 22: number analyzed (Participants) | 15 | 25 | 38
  Week 22 | -138.67 (147.069) | -125.18 (165.395) | -73.24 (126.319)
  Week 24: number analyzed (Participants) | 14 | 30 | 50
  Week 24 | -112.96 (175.107) | -133.52 (191.550) | -65.37 (128.580)
  Weeks 36: number analyzed (Participants) | 17 | 29 | 49
  Weeks 36 | -129.41 (179.357) | -114.19 (200.789) | -60.90 (128.520)
  Week 46: number analyzed (Participants) | 11 | 25 | 38
  Week 46 | -166.05 (195.963) | -156.88 (157.687) | -63.80 (128.199)
  Week 48: number analyzed (Participants) | 13 | 26 | 45
  Week 48 | -145.65 (177.520) | -121.73 (114.214) | -57.90 (143.238)
  Week 60: number analyzed (Participants) | 13 | 27 | 47
  Week 60 | -86.46 (159.360) | -133.17 (162.933) | -43.31 (125.923)
  Week 70: number analyzed (Participants) | 10 | 23 | 33
  Week 70 | -149.02 (186.918) | -146.43 (196.501) | -50.08 (140.232)
  Week 72: number analyzed (Participants) | 13 | 26 | 40
  Week 72 | -101.31 (169.631) | -123.44 (143.220) | -52.39 (156.473)

5. Secondary Outcome: Proportion of Positive Pruritus Assessments at the Participant Level Using the Albireo ObsRo Instrument From Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 34-36, 44-46, 47-48, 58-60, 68-70, 71-72, 73-76
Description: as for outcome 2
Time Frame: Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 34-36, 44-46, 47-48, 58-60, 68-70, 71-72, 73-76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of pruritus-participant-level
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 37 | 53
proportion of pruritus-participant-level
  Weeks 1-4 | 45.72 (34.300) | 23.64 (27.005) | 60.14 (33.985)
  Weeks 5-8: number analyzed (Participants) | 19 | 37 | 51
  Weeks 5-8 | 53.75 (39.894) | 28.76 (32.349) | 71.14 (34.866)
  Weeks 9-12: number analyzed (Participants) | 19 | 37 | 50
  Weeks 9-12 | 54.01 (41.345) | 29.64 (35.594) | 71.03 (36.961)
  Weeks 13-16: number analyzed (Participants) | 18 | 37 | 50
  Weeks 13-16 | 57.47 (42.420) | 31.78 (36.364) | 72.19 (39.221)
  Weeks 17-20: number analyzed (Participants) | 18 | 36 | 48
  Weeks 17-20 | 55.28 (41.441) | 36.15 (38.564) | 73.95 (38.051)
  Weeks 21-24: number analyzed (Participants) | 17 | 36 | 45
  Weeks 21-24 | 55.62 (42.927) | 35.83 (40.132) | 73.11 (37.875)
  Weeks 34-36: number analyzed (Participants) | 16 | 31 | 43
  Weeks 34-36 | 58.24 (41.117) | 32.79 (39.066) | 72.39 (35.581)
  Weeks 44-46: number analyzed (Participants) | 14 | 28 | 37
  Weeks 44-46 | 67.33 (39.242) | 38.40 (43.144) | 77.11 (31.712)
  Weeks 47-48: number analyzed (Participants) | 14 | 29 | 41
  Weeks 47-48 | 67.31 (43.702) | 34.71 (42.594) | 71.86 (39.020)
  Weeks 58-60: number analyzed (Participants) | 13 | 31 | 35
  Weeks 58-60 | 65.82 (40.745) | 44.22 (43.534) | 72.31 (38.008)
  Weeks 68-70: number analyzed (Participants) | 13 | 22 | 29
  Weeks 68-70 | 62.43 (40.321) | 56.79 (42.935) | 69.40 (39.034)
  Weeks 71-72: number analyzed (Participants) | 12 | 26 | 31
  Weeks 71-72 | 57.65 (39.797) | 55.75 (45.076) | 72.26 (38.680)
  Weeks 73-76: number analyzed (Participants) | 3 | 8 | 9
  Weeks 73-76 | 41.59 (39.923) | 63.48 (29.003) | 69.23 (33.797)

6. Secondary Outcome: Proportion of Positive Pruritus Assessments at the Participant Level Using the Albireo ObsRo Instrument (AM Score)
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least a 1-point drop from baseline on the Albireo ObsRO instrument. The proportion of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant. AM score represents night-time itching/scratching and sleep disturbance.
Time Frame: Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 34-36, 44-46, 47-48, 58-60, 68-70, 71-72, and 73-76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of pruritus-participant-level
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 36 | 53
proportion of pruritus-participant-level
  Weeks 1-4 | 42.38 (36.177) | 23.72 (29.373) | 58.19 (36.799)
  Weeks 5-8: number analyzed (Participants) | 19 | 36 | 51
  Weeks 5-8 | 48.16 (42.655) | 27.70 (34.144) | 69.00 (38.199)
  Weeks 9-12: number analyzed (Participants) | 19 | 36 | 49
  Weeks 9-12 | 50.57 (42.880) | 28.41 (37.802) | 68.96 (38.876)
  Weeks 13-16: number analyzed (Participants) | 18 | 36 | 48
  Weeks 13-16 | 53.47 (43.689) | 31.70 (38.438) | 69.03 (41.902)
  Weeks 17-20: number analyzed (Participants) | 18 | 36 | 47
  Weeks 17-20 | 53.94 (42.837) | 35.37 (40.673) | 71.30 (40.934)
  Weeks 21-24: number analyzed (Participants) | 17 | 36 | 45
  Weeks 21-24 | 55.52 (44.798) | 35.15 (41.940) | 69.63 (40.353)
  Weeks 34-36: number analyzed (Participants) | 16 | 29 | 43
  Weeks 34-36 | 57.49 (43.512) | 34.80 (39.644) | 69.92 (37.610)
  Weeks 44-46: number analyzed (Participants) | 14 | 27 | 36
  Weeks 44-46 | 67.07 (42.321) | 40.11 (43.580) | 73.62 (37.122)
  Weeks 47-48: number analyzed (Participants) | 14 | 28 | 41
  Weeks 47-48 | 63.67 (46.870) | 35.60 (42.748) | 69.18 (42.923)
  Weeks 58-60: number analyzed (Participants) | 13 | 30 | 33
  Weeks 58-60 | 59.54 (45.249) | 46.44 (44.871) | 70.83 (40.675)
  Weeks 68-70: number analyzed (Participants) | 13 | 21 | 28
  Weeks 68-70 | 62.42 (42.359) | 63.21 (43.450) | 64.35 (44.147)
  Weeks 71-72: number analyzed (Participants) | 12 | 27 | 30
  Weeks 71-72 | 60.18 (41.743) | 60.74 (43.254) | 71.45 (41.406)
  Weeks 73-76: number analyzed (Participants) | 3 | 8 | 10
  Weeks 73-76 | 33.22 (52.059) | 62.66 (29.530) | 69.93 (36.023)

7. Secondary Outcome: Proportion of Positive Pruritus Assessments at the Participant Level Using the Albireo ObsRo Instrument (PM Score)
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least a 1-point drop from baseline on the Albireo ObsRO instrument. The proportion of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant. PM score represents daytime itching/scratching and tiredness.
Time Frame: Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 34-36, 44-46, 47-48, 58-60, 68-70, 71-72, and 73-76
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of pruritus-participant-level
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 37 | 53
proportion of pruritus-participant-level
  Weeks 1-4 | 49.01 (35.687) | 24.13 (30.344) | 62.08 (34.404)
  Weeks 5-8: number analyzed (Participants) | 19 | 37 | 51
  Weeks 5-8 | 60.03 (39.300) | 30.45 (35.987) | 73.11 (36.284)
  Weeks 9-12: number analyzed (Participants) | 19 | 37 | 50
  Weeks 9-12 | 57.77 (42.435) | 31.73 (38.223) | 72.42 (37.687)
  Weeks 13-16: number analyzed (Participants) | 18 | 37 | 50
  Weeks 13-16 | 61.36 (41.530) | 33.08 (39.999) | 74.13 (38.607)
  Weeks 17-20: number analyzed (Participants) | 18 | 37 | 48
  Weeks 17-20 | 56.49 (41.590) | 36.22 (41.689) | 76.12 (36.907)
  Weeks 21-24: number analyzed (Participants) | 17 | 36 | 46
  Weeks 21-24 | 55.78 (43.495) | 36.28 (41.318) | 77.23 (37.626)
  Weeks 34-36: number analyzed (Participants) | 16 | 31 | 43
  Weeks 34-36 | 58.75 (39.774) | 30.28 (39.297) | 75.11 (36.650)
  Weeks 44-46: number analyzed (Participants) | 14 | 28 | 37
  Weeks 44-46 | 67.01 (39.601) | 38.02 (43.252) | 81.00 (30.974)
  Weeks 47-48: number analyzed (Participants) | 14 | 29 | 41
  Weeks 47-48 | 71.08 (41.878) | 34.98 (43.148) | 74.62 (38.856)
  Weeks 58-60: number analyzed (Participants) | 13 | 31 | 33
  Weeks 58-60 | 72.28 (38.149) | 43.53 (43.694) | 73.17 (38.473)
  Weeks 68-70: number analyzed (Participants) | 13 | 21 | 28
  Weeks 68-70 | 62.63 (40.626) | 55.65 (42.883) | 74.85 (38.702)
  Weeks 71-72: number analyzed (Participants) | 12 | 26 | 32
  Weeks 71-72 | 55.12 (42.336) | 53.97 (45.611) | 75.38 (39.038)
  Weeks 73-76: number analyzed (Participants) | 3 | 8 | 10
  Weeks 73-76 | 49.36 (36.671) | 63.35 (31.538) | 68.11 (32.377)

8. Secondary Outcome: Percentage of Responders for Pruritus Assessments Bi-Weekly (AM and PM)
Description: A responder is defined as a participant who reports a decrease in pruritus score from unrounded baseline equivalent to or greater than the threshold of meaningful change estimated from the blinded psychometric analysis. The averaged pruritus score was used to calculate the percentage of participants achieving meaningful reduction at specified Week against the thresholds value of 1.00 based on bi-weekly scores at specified Week obtained from blinded psychometric analysis across all anchors support a threshold of 1.0 point for AM, PM and AM and PM scratching scores. ObsRO instrument was used to assess severity of observed scratching twice a day (AM and PM) with score from 0 to 4 where 0 is no scratching and 4 is worst possible scratching.
Time Frame: Weeks 1-2, 3-4, 5-6, 7-8, 9-10, 11-12, 13-14, 15-16, 17-18, 19-20, 21-22, 23-24, 35-36, 47-48, 59-60, and 71-72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 36 | 53
percentage of participants
  Weeks 1-2 | 15.8 [3.38 to 39.58] | 2.8 [0.07 to 14.53] | 28.3 [16.79 to 42.35]
  Weeks 3-4 | 36.8 [16.29 to 61.64] | 2.8 [0.07 to 14.53] | 52.8 [38.64 to 66.70]
  Weeks 5-6: number analyzed (Participants) | 19 | 36 | 52
  Weeks 5-6 | 36.8 [16.29 to 61.64] | 5.6 [0.68 to 18.66] | 55.8 [41.33 to 69.53]
  Weeks 7-8: number analyzed (Participants) | 19 | 36 | 51
  Weeks 7-8 | 36.8 [16.29 to 61.64] | 13.9 [4.67 to 29.50] | 54.9 [40.34 to 68.87]
  Weeks 9-10: number analyzed (Participants) | 19 | 36 | 50
  Weeks 9-10 | 31.6 [12.58 to 56.55] | 8.3 [1.75 to 22.47] | 58.0 [43.21 to 71.81]
  Weeks 11-12: number analyzed (Participants) | 18 | 36 | 50
  Weeks 11-12 | 33.3 [13.34 to 59.01] | 13.9 [4.67 to 29.50] | 56.0 [41.25 to 70.01]
  Weeks 13-14: number analyzed (Participants) | 18 | 36 | 50
  Weeks 13-14 | 50.0 [26.02 to 73.98] | 11.1 [3.11 to 26.06] | 58.0 [43.21 to 71.81]
  Weeks 15-16: number analyzed (Participants) | 18 | 36 | 49
  Weeks 15-16 | 50.0 [26.02 to 73.98] | 13.9 [4.67 to 29.50] | 57.1 [42.21 to 71.18]
  Weeks 17-18: number analyzed (Participants) | 18 | 36 | 47
  Weeks 17-18 | 44.4 [21.53 to 69.24] | 16.7 [6.37 to 32.81] | 55.3 [40.12 to 69.83]
  Weeks 19-20: number analyzed (Participants) | 16 | 36 | 48
  Weeks 19-20 | 50.0 [24.65 to 75.35] | 22.2 [10.12 to 39.15] | 56.3 [41.18 to 70.52]
  Weeks 21-22: number analyzed (Participants) | 17 | 36 | 45
  Weeks 21-22 | 41.2 [18.44 to 67.08] | 16.7 [6.37 to 32.81] | 57.8 [42.15 to 72.34]
  Weeks 23-24: number analyzed (Participants) | 17 | 36 | 46
  Weeks 23-24 | 41.2 [18.44 to 67.08] | 19.4 [8.19 to 36.02] | 56.5 [41.11 to 71.07]
  Weeks 35-36: number analyzed (Participants) | 15 | 27 | 39
  Weeks 35-36 | 33.3 [11.82 to 61.62] | 18.5 [6.30 to 38.08] | 56.4 [39.62 to 72.19]
  Weeks 47-48: number analyzed (Participants) | 14 | 28 | 39
  Weeks 47-48 | 57.1 [28.86 to 82.34] | 25.0 [10.69 to 44.87] | 64.1 [47.18 to 78.80]
  Weeks 59-60: number analyzed (Participants) | 11 | 30 | 30
  Weeks 59-60 | 36.4 [10.93 to 69.21] | 30.0 [14.73 to 49.40] | 60.0 [40.60 to 77.34]
  Weeks 71-72: number analyzed (Participants) | 12 | 26 | 31
  Weeks 71-72 | 41.7 [15.17 to 72.33] | 34.6 [17.21 to 55.67] | 61.3 [42.19 to 78.15]

9. Secondary Outcome: Percentage of Responders for Pruritus Assessments Monthly (AM and PM)
Description: A responder is defined as a participant who reports a decrease in pruritus score from unrounded baseline equivalent to or greater than the threshold of meaningful change estimated from the blinded psychometric analysis. The averaged pruritus score was used to calculate the percentage of participants achieving meaningful reduction at specified Week against the thresholds value of 1.00 based on monthly scores at specified Week obtained from blinded psychometric analysis across all anchors support a threshold of 1.0 point for AM, PM and AM and PM scratching scores. ObsRO instrument was used to assess severity of observed scratching twice a day (AM and PM) with score from 0 to 4 where 0 is no scratching and 4 is worst possible scratching.
Time Frame: Weeks 1-4, 5-8, 9-12, 13-16, 17-20, 21-24, 34-36, 45-48, 58-60, and 68-72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 36 | 53
percentage of participants
  Weeks 1-4 | 21.1 [6.05 to 45.57] | 2.8 [0.07 to 14.53] | 43.4 [29.84 to 57.72]
  Weeks 5-8: number analyzed (Participants) | 19 | 36 | 51
  Weeks 5-8 | 36.8 [16.29 to 61.64] | 8.3 [1.75 to 22.47] | 54.9 [40.34 to 68.87]
  Weeks 9-12: number analyzed (Participants) | 19 | 36 | 50
  Weeks 9-12 | 36.8 [16.29 to 61.64] | 11.1 [3.11 to 26.06] | 56.0 [41.25 to 70.01]
  Weeks 13-16: number analyzed (Participants) | 18 | 36 | 50
  Weeks 13-16 | 50.0 [26.02 to 73.98] | 13.9 [4.67 to 29.50] | 60.0 [45.18 to 73.59]
  Weeks 17-20: number analyzed (Participants) | 18 | 36 | 48
  Weeks 17-20 | 38.9 [17.30 to 64.25] | 16.7 [6.37 to 32.81] | 56.3 [41.18 to 70.52]
  Weeks 21-24: number analyzed (Participants) | 17 | 36 | 45
  Weeks 21-24 | 35.3 [14.21 to 61.67] | 16.7 [6.37 to 32.81] | 53.3 [37.87 to 68.34]
  Weeks 34-36: number analyzed (Participants) | 16 | 30 | 43
  Weeks 34-36 | 43.8 [19.75 to 70.12] | 23.3 [9.93 to 42.28] | 58.1 [42.13 to 72.99]
  Weeks 45-48: number analyzed (Participants) | 15 | 29 | 39
  Weeks 45-48 | 53.3 [26.59 to 78.73] | 24.1 [10.30 to 43.54] | 64.1 [47.18 to 78.80]
  Weeks 58-60: number analyzed (Participants) | 13 | 31 | 35
  Weeks 58-60 | 46.2 [19.22 to 74.87] | 29.0 [14.22 to 48.04] | 57.1 [39.35 to 73.68]
  Weeks 68-72: number analyzed (Participants) | 13 | 24 | 31
  Weeks 68-72 | 53.8 [25.13 to 80.78] | 37.5 [18.80 to 59.41] | 64.5 [45.37 to 80.77]

10. Secondary Outcome: Percentage of Participants Achieving a Positive Pruritus Assessment for >50% of the Time Based on the Albireo ObsRO (AM and PM)
Description: The percentage of participants who achieved positive pruritus assessment for more than 50% of the time for Weeks 0-72 is reported. A positive pruritus assessment is defined as a scratching score of <=1 or at least a 1-point decrease from baseline on the Albireo ObsRO instrument based on rounded baseline and was calculated based on reported eDiary data. At each assessment, the AM score was compared to the baseline AM average, and the PM score was compared to the baseline PM average. All assessments after intercurrent events (premature treatment discontinuation, death, or initiation of rescue treatments such as biliary diversion surgery or liver transplantation) or follow-up assessments (>= last dose day + 15 days) were excluded from analysis.
Time Frame: Week 72
Population: The FAS consisted of all participants who had received at least 1 dose of the study treatment. Only participants with non-missing value when >50% were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 12 | 26 | 31
percentage of participants | 58.3 [27.67 to 84.83] | 34.6 [17.21 to 55.67] | 83.9 [66.27 to 94.55]

11. Secondary Outcome: Number of Participants Who Underwent Biliary Diversion Surgery and Liver Transplantation
Description: Participants who underwent biliary diversion surgery and or liver transplantation data has been reported.
Time Frame: Baseline and Weeks 24, 48, and 72
Population: The FAS consisted of all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 37 | 60
Participants
  Weeks 0-24: Biliary Diversion Surgery | 0 | 0 | 0
  Weeks 0-24: Liver Transplantation | 1 | 0 | 0
  Weeks 0-48: Biliary Diversion Surgery | 1 | 0 | 1
  Weeks 0-48: Liver Transplantation | 2 | 0 | 2
  Weeks 0-72: Biliary Diversion Surgery | 1 | 0 | 1
  Weeks 0-72: Liver Transplantation | 2 | 0 | 5

12. Secondary Outcome: Change From Baseline in Height Z-Scores
Description: Growth factors like height was measured by the standardized assessments outlined in the US food and drug administration (FDA) guidance document. Height was measured using certified stadiometer. Change in growth parameters was assessed using linear growth (height) compared to standard growth curve (Z-score) calculated by using the software or methods from the centers for disease control (CDC) website for participants with age >=2 years old and from the world health organization (WHO) website for participants with age <2 years old. Participants whose accurate age was not available, Z-score was not calculated. Baseline is the last available assessment prior to first dose of study treatment. A Z-score indicates how many standard deviation's (SD) a participant's measurement (like height), was from the average for their age and sex. A Z-score of 0 represents the median or 50th percentile, while positive or negative values show how far above or below average a measurement was.
Time Frame: Baseline and Weeks 24, 48, 70 and 72
Population: as for outcome 1
Measure: Median (Full Range); unit: Z-score
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 15 | 28 | 46
Z-score
  Week 24: number analyzed (Participants) | 14 | 28 | 46
  Week 24 | 0.181 [-0.28 to 1.53] | 0.341 [-1.04 to 2.26] | 0.089 [-1.34 to 1.97]
  Week 48: number analyzed (Participants) | 14 | 27 | 41
  Week 48 | 0.485 [0.02 to 1.42] | 0.662 [-0.75 to 2.08] | 0.095 [-1.46 to 2.03]
  Average of Weeks 70-72: number analyzed (Participants) | 15 | 28 | 39
  Average of Weeks 70-72 | 0.556 [-0.01 to 1.57] | 0.543 [-0.83 to 2.12] | 0.224 [-1.42 to 2.62]

13. Secondary Outcome: Change From Baseline in Weight Z-Scores
Description: Growth factors like weight was measured by the standardized assessments outlined in the US FDA guidance document. Weight was measured using certified weight scale. Change in growth parameters was assessed using linear growth (weight) compared to standard growth curve (Z-score), calculated by using the software or methods from the CDC website for participants with age >=2 years old and from the WHO website for participants with age <2 years old. Participants whose accurate age was not available, Z-score was not calculated. Baseline is the last available assessment prior to the first dose of study treatment. The Z-score indicates how many SDs a participant's measurement (like weight), was from the average for their age and sex. A Z-score of 0 represents the median or 50th percentile, while positive or negative values show how far above or below the average a measurement was.
Time Frame: Baseline and Weeks 24, 48, 70 and 72
Population: as for outcome 1
Measure: Median (Full Range); unit: Z-score
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 15 | 29 | 48
Z-score
  Week 24: number analyzed (Participants) | 14 | 29 | 48
  Week 24 | 0.155 [-0.49 to 1.40] | 0.383 [-0.75 to 1.57] | 0.169 [-0.68 to 1.74]
  Week 48: number analyzed (Participants) | 14 | 27 | 42
  Week 48 | 0.544 [-1.15 to 1.43] | 0.494 [-1.04 to 2.14] | 0.246 [-0.54 to 1.29]
  Average of Weeks 70-72: number analyzed (Participants) | 15 | 28 | 40
  Average of Weeks 70-72 | 0.098 [-1.13 to 2.17] | 0.389 [-1.21 to 2.11] | 0.400 [-0.86 to 2.27]

14. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Z-Scores
Description: Growth factors like BMI was measured by the standardized assessments outlined in the US FDA guidance document. BMI was calculated by weight (kg) / height (m)^2. Change in growth parameters was assessed using linear growth (BMI) compared to standard growth curve (Z-score), calculated by using the software or methods from the CDC website for participants with age >=2 years old and from the WHO website for participants with age <2 years old. Participants whose accurate age was not available, Z-score was not calculated. Baseline is the last available assessment prior to the first dose of study treatment. The Z-score indicates how many SDs a participant's measurement (like BMI), was from the average for their age and sex. A Z-score of 0 represents the median or 50th percentile, while positive or negative values show how far above or below the average a measurement was.
Time Frame: Baseline and Weeks 24, 48, 70 and 72
Population: as for outcome 1
Measure: Median (Full Range); unit: Z-score
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 15 | 28 | 46
Z-score
  Week 24: number analyzed (Participants) | 14 | 28 | 46
  Week 24 | -0.106 [-0.66 to 1.86] | 0.150 [-2.00 to 2.21] | 0.202 [-1.60 to 2.08]
  Week 48: number analyzed (Participants) | 14 | 27 | 41
  Week 48 | 0.028 [-0.88 to 1.23] | -0.135 [-2.44 to 2.59] | 0.129 [-1.34 to 2.45]
  Average of Weeks 70-72: number analyzed (Participants) | 15 | 28 | 39
  Average of Weeks 70-72 | -0.059 [-1.24 to 3.12] | -0.007 [-1.64 to 2.25] | 0.182 [-0.99 to 2.68]

15. Secondary Outcome: Number of Participants With Use of Ursodeoxycholic Acid (UDCA) and/or Rifampicin at Weeks 24, 48, and 72
Description: Data for the number of participants with use of UDCA and rifampicin are reported.
Time Frame: Weeks 24, 48, and 72
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 19 | 37 | 60
Participants
  Week 24: Use of UDCA | 17 | 29 | 43
  Week 24: Use of Rifampicin | 17 | 19 | 37
  Week 24: Use of UDCA or Rifampicin | 19 | 33 | 50
  Week 24: Use of UDCA and Rifampicin | 15 | 15 | 30
  Week 48: Use of UDCA: number analyzed (Participants) | 18 | 35 | 56
  Week 48: Use of UDCA | 16 | 27 | 39
  Week 48: Use of Rifampicin: number analyzed (Participants) | 18 | 35 | 56
  Week 48: Use of Rifampicin | 16 | 20 | 31
  Week 48: Use of UDCA or Rifampicin: number analyzed (Participants) | 18 | 35 | 56
  Week 48: Use of UDCA or Rifampicin | 18 | 33 | 46
  Week 48: Use of UDCA and Rifampicin: number analyzed (Participants) | 18 | 35 | 56
  Week 48: Use of UDCA and Rifampicin | 14 | 14 | 24
  Week 72: Use of UDCA: number analyzed (Participants) | 16 | 31 | 50
  Week 72: Use of UDCA | 14 | 24 | 34
  Week 72: Use of Rifampicin: number analyzed (Participants) | 16 | 31 | 50
  Week 72: Use of Rifampicin | 14 | 15 | 26
  Week 72: Use of UDCA or Rifampicin: number analyzed (Participants) | 16 | 31 | 50
  Week 72: Use of UDCA or Rifampicin | 16 | 29 | 41
  Week 72: Use of UDCA and Rifampicin: number analyzed (Participants) | 16 | 31 | 50
  Week 72: Use of UDCA and Rifampicin | 12 | 10 | 19

16. Secondary Outcome: Change From Baseline to Week 72 in Pediatric End-Stage Liver Disease (PELD) Score
Description: The PELD score was calculated for children under 12 years of age, ranged across negative to positive values. The calculation of the PELD score was done by converting the laboratory parameters: total bilirubin in milligram/deciliter (mg/dL), albumin in gram (g)/dL, and creatinine in mg/dL laboratory parameters were converted to units. PELD score was calculated as 4.80*ln (total bilirubin)+18.57*ln [international normalized ratio (INR)] - 6.87*ln (albumin) + 4.36 (if participant <1 year: scores for participants listed for liver transplantation before the participant's first birthday continued to include the value assigned for age (<1 year) until the participant reached the age of 24 months) + 6.67 (if the participant has growth failure [<-2 standard deviation]). The laboratory values <1.0 were set to 1.0 for the calculation of the PELD score. Lower scores represent less severe hepatic disease. Baseline is the last available assessment prior to the first dose of study treatment.
Time Frame: Baseline and Week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 11 | 20 | 23
score on a scale | -0.397 (3.6168) | 1.361 (2.5083) | -0.303 (9.4631)

17. Secondary Outcome: Change From Baseline to Week 72 in Model for End-stage Liver Disease (MELD) Score for Children 12 Years of Age or Older
Description: The MELD score was calculated for children 12 years of age or older ranges from 6 to 40. The calculation of the MELD score was done by converting the laboratory parameters in the following units: total bilirubin in mg/dL, albumin in g/dL, and creatinine in mg/dL laboratory parameters were converted to units. MELD score for children 12 years of age or older ranges from 6 to 40 was calculated as 9.57*ln (creatinine) + 3.78*ln (total bilirubin) + 11.2 *ln (INR) + 6.43. Laboratory values <1.0 were set to 1.0 and serum creatinine values >4.0 mg/dL were set to 4.0 for calculation of the MELD score. Lower scores represent less severe hepatic disease. Baseline is the last available assessment prior to the first dose of study treatment.
Time Frame: Baseline and Week 72
Population: The FAS consisted of all participants who had received at least 1 dose of the study treatment. Only participants 12 years of age or older are included in this analysis and reported. For Cohort 1: Placebo/Odevixibat change from baseline data was not collected as participant was under 12 years old, that aligns with MELD score calculation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 1 | 3 | 17
score on a scale
  Baseline | 6.869 (NA) — NA indicates standard deviation not calculated for single participant. | 9.795 (2.4694) | 11.574 (4.0801)
  Change from Baseline: number analyzed (Participants) | 0 | 1 | 9
  Change from Baseline |  | 1.286 (NA) — NA indicates standard deviation not calculated for single participant. | -2.221 (5.7744)

18. Secondary Outcome: Change From Baseline to Week 72 in Aspartate Aminotransferase (AST) to Platelet Ratio Index (APRI) Score
Description: AST to APRI score was calculated as [(AST in units per liter {U/L})/ (AST upper limit of normal {ULN} in U/L)] * 100/ (platelets in 10^9/L). The APRI score is a way to assess fibrosis of the liver. The lower the APRI score (< 0.5), the greater the negative predictive value and ability to rule out cirrhosis; the higher the value (> 1.5) the greater the positive predictive value and ability to rule in cirrhosis. Lower values indicate less severe hepatic fibrosis. Baseline is the last available assessment prior to the first dose of study treatment.
Time Frame: Baseline and Week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 13 | 21 | 22
score on a scale | 0.044 (0.3435) | 0.071 (0.3951) | 0.411 (0.9690)

19. Secondary Outcome: Change From Baseline to Week 72 in Fibrosis-4 (Fib-4) Score
Description: Fib-4 score was calculated as (age * AST in U/L)/ (platelets in 10^9/L *√ ( alanine aminotransferase [ALT] in U/L). The FIB-4 score estimates the amount of scarring in the liver. A FIB-4 score <1.45 has a negative predictive value of 90% for advanced fibrosis (Ishak fibrosis score 4-6 which includes early bridging fibrosis to cirrhosis). In contrast, a FIB-4 > 3.25 would have a 97% specificity and a positive predictive value of 65% for advanced fibrosis. Lower values indicate less severe hepatic fibrosis. Baseline is the last available assessment prior to the first dose of study treatment.
Time Frame: Baseline and Week 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
Number analyzed (Participants) | 13 | 21 | 21
score on a scale | 0.050 (0.1187) | 0.106 (0.2696) | 0.113 (0.2820)

ADVERSE EVENTS:
Time Frame: Treatment emergent serious adverse event (TESAEs) and non-serious treatment emergent adverse event (TEAEs) were collected from the start of study treatment administration (Day 1) up to 28 days after the last dose of study treatment, approximately 248 weeks. All-cause mortality (death) was assessed from signing of the informed consent form till DCO, approximately 281 weeks.
Description: The FAS consisted of all participants who had received at least 1 dose of the study treatment.
Arm/Group | Cohort 1: Placebo/Odevixibat | Cohort 1: Odevixibat/Odevixibat | Cohort 2: Odevixibat
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/37 | 0/60
Serious Adverse Events (participants affected / at risk) | 5/19 | 7/37 | 23/60
Other Adverse Events (participants affected / at risk) | 18/19 | 35/37 | 57/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo/Odevixibat (N=19) | Cohort 1: Odevixibat/Odevixibat (N=37) | Cohort 2: Odevixibat (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Progressive familial intrahepatic cholestasis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (3)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic arthritis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alpha 1 foetoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo/Odevixibat (N=19) | Cohort 1: Odevixibat/Odevixibat (N=37) | Cohort 2: Odevixibat (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 4 (4)
Ear discomfort (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (3) | 3 (3) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 2 (4) | 0 (0)
Keratoconus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (6) | 4 (4)
Dental caries (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 8 (16) | 16 (20)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 10 (15)
Pyrexia (General disorders) | 7 (17) | 12 (25) | 16 (29)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 4 (4) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2) | 3 (3)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Boston exanthema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (4) | 2 (4)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3) | 15 (17)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 2 (4) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (2) | 5 (5) | 6 (6)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 7 (10) | 8 (11)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 9 (16) | 9 (10)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 2 (3) | 3 (9) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (4)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 3 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (4) | 3 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (21) | 10 (19) | 12 (17)
Varicella (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 1 (2) | 4 (5) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post vaccination fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 5 (10)
Bile acids increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 3 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (6) | 10 (17) | 13 (20)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood sodium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 3 (3) | 5 (7) | 11 (13)
Lymph node palpable (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 2 (2) | 3 (4)
Vitamin A increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 2 (4) | 2 (2)
Vitamin E decreased (Investigations) | 1 (2) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 8 (9)
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 13 (23) | 10 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (5) | 6 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (3) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (10) | 7 (8)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT03659916/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT03659916/SAP_001.pdf